CLINICAL TRIAL: NCT07090356
Title: Effects of Instrument-Assisted Soft Tissue Mobilization Versus Proprioceptive Neuromuscular Facilitation Stretching in Athletes With Piriformis Syndrome
Brief Title: Instrument-Assisted Soft Tissue Mobilization Versus PNF Stretching in Athletes With Piriformis Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0460
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assesor Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument-Assisted Soft Tissue Mobilization (Experimental): IASTM therapy will be provided to participants in whom a specialized instrument wwill be used to apply controlled pressure over the piriformis muscle as well as surrounding soft tissues.
  Interventions: Other: Instrument-Assisted Soft Tissue Mobilization
- Proprioceptive Neuromuscular Facilitation Stretching (Experimental): PNF stretching (contract relax; hold relax) was implemented to stretch participants' muscles as flexibly and with as much control as possible.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation Stretching

INTERVENTIONS:
Other: Instrument-Assisted Soft Tissue Mobilization — IASTM therapy will be provided to participants in whom a specialized instrument will be used to apply controlled pressure over the piriformis muscle as well as surrounding soft tissues.
  Arms: Instrument-Assisted Soft Tissue Mobilization
Other: Proprioceptive Neuromuscular Facilitation Stretching — PNF stretching (contract relax; hold relax) will be implemented to stretch participants' muscles as flexibly and with as much control as possible.
  Arms: Proprioceptive Neuromuscular Facilitation Stretching

SUMMARY:
A 12-month randomized controlled trial will be conducted at Pakistan Sports Board, Lahore, with 40 athletes (18-35 years) randomly allocated to IASTM (n=20) or PNF (n=20) groups. Interventions were administered 3 times/week for 4 weeks. Outcomes included Numeric Pain Rating Scale (NPRS), goniometric hip ROM, and Oswestry Disability Index (ODI).

DETAILED DESCRIPTION:
The objective of this study will be to compare the effectiveness of IASTM versus PNF stretching to manage Piriformis Syndrome in a 4 - week randomized controlled trial (RCT). Random allocation was done to the IASTM group or the PNF stretching group. Physiotherapy interventions to reduce pain, increase muscle flexibility and increase functional outcomes will be given to both groups.

Before the intervention, all participants will underween a comprehensive assessment, including:

* Numeric Pain Rating Scale (NPRS) for pain intensity
* Oswestry Disability Index (ODI) for functional disability
* Goniometric measurement for hip joint range of motion (ROM)

Group A: Instrument-Assisted Soft Tissue Mobilization (IASTM) Group

IASTM therapy was provided to participants in whom a specialized instrument was used to apply controlled pressure over the piriformis muscle as well as surrounding soft tissues. The procedure included:

* Warm-up: Light aerobic exercise (5 minutes)
* IASTM Application: Applied over the piriformis muscle in a longitudinal and cross-fiber pattern for 5-7 minutes
* Static stretching of the piriformis and gluteal muscle activation exercises are completed next.
* Cool-down: Light stretching and relaxation

Group B: Proprioceptive Neuromuscular Facilitation (PNF) Stretching Group

PNF stretching (contract relax; hold relax) was implemented to stretch participants' muscles as flexibly and with as much control as possible. The procedure included:

* Warm-up: Light aerobic exercise (5 minutes)
* PNF Stretching:

  * The second technique was based on hold-relax technique during which the participant actively contracted the piriformis muscle against resistance for 5 seconds, followed by a 10 seconds passive stretch.
  * Contract relax technique: same as the above but with deeper stretches following an active contraction
  * Repeated for 3 sets per session
* Exercises to strengthen the core and hip muscles to provide stability
* Gentle stretching and deep breathing for cool down

Physiotherapy Management (Common for Both Groups)

In addition, the following was provided to all the participants together with their respective interventions:

* Ice/heat application as needed (based on the individual).
* Education & Ergonomic Advice: Guidance on proper posture, activity modification, and self-care techniques Specific exercises will be assigned to maintain flexibility and strength (Home Exercise Program).

ELIGIBILITY:
Inclusion Criteria:

* Professional Athletes aged 18 to 35 years.
* Chronic pain in the buttock and hip area.
* Inability to sit for a prolonged time.
* Athletes having positive Faber test
* Both male and female athletes
* Practicing athletes who are in practice from last 2 years.

Exclusion Criteria:

* Trauma history from last 6 months.
* Other injuries excluding hip pain.
* Systemic illness.
* Pre-existing neurological conditions affecting the lower limbs
* History of lower back surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  Numeric Pain Rating Scale
Hip ROM | 6 weeks
  Goniometry
Oswestry Disability Index | 6 weeks
  Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No